CLINICAL TRIAL: NCT04987372
Title: Comparison of Pain and Comfort in Patients Following Cardiac Surgery: Opioid- Morphine Managed Versus Multimodal Pain-management
Brief Title: Multimodal Versus Opioid aNalgesia in carDiAc Surgery
Acronym: MONDAY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-000515-84
Record Dates: First submitted 2019-08-14; First posted 2021-08-03 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Pain; Postoperative Delirium
MeSH Terms: conditions — Pain, Postoperative; Emergence Delirium | interventions — Dexmedetomidine; Ketamine; Lidocaine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Classical protocol (No Intervention): Fentanyl Max. 15µg/kg IV Per-operative
  Ultiva (Remifentanyl) 0.02-0.1µg/kg/h IV Post-operative
  Paracetamol 4x1g /24h IV Post-operative
  Tradonal (Tramadol) 100mg IV 4/d IV Post-operative in cas of break through pain
  Oxynorm (Oxycodon) 5-10mg 4-6/d PO Post-operative in case of Break through pain
- Multimodal protocol (Active Comparator): Lyrica (Pregabalin) 75mg PO 2 hours before the operation
  Dexdor (Dexmedetomidine) 0.8µg/kg/h IV Per-operative / Post-operative
  Ketalar (Ketamine) Bolus (0.5mg/kg) + 0.3mg/kg/h IV Per-operative until stop propofol
  Linisol (Lidocain) Bolus (1.5mg/kg) + 1.3mg/kg/h IV Per-operatiive until 12h post-op
  Magnesium Sulphate Induction (25mg/kg) + 25mg/kg weaning ECC IV Per-operative
  Fentanyl 2.5µg/kg IV Per-operative
  Paracetamol 4x1g /24u IV Post-operative
  Tradonal (Tramadol) 100mg IV 4/d IV Post-operative in case of Break through pain
  Oxynorm (Oxycodon) 5-10mg 4-6/d PO Post-operative in case of Break through pain
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The use of multimodal painkillers pre, per and postoperative
  Other Names: pregabaline; ketamine; lidocaine; magnesium sulfate
  Arms: Multimodal protocol

SUMMARY:
To compare standard "Fentanyl - Tramadol - Paracetamol - Oxycodone" regimen to a multimodal painmanagement "pregabalin- minimal fentanyl-ketamine-lidocain-dexmedetomidine- paracetamol" to determine which therapy provides the most comfort, the fastest extubation time, the least pain and the least delirium.

DETAILED DESCRIPTION:
Cardiac surgery for the adult, performed by sternotomy is associated with moderate to severe acute postoperative pain. Postoperative pain is the primary reason for prolonged convalescence and one of the main concerns of the surgical patient in the Intensive Care Unit (ICU). This pain is multifactorial and multifocal; and can be caused by incision, intraoperative tissue retraction and dissection, surgical manipulation of the parietal pleura, posterior rib dislocation or fracture, possible brachial plexus injury, chest tube insertion and harvesting of the saphenous vein and internal mammarian artery.

The most common analgesic schemes for postoperative pain in cardiac surgery are based on intravenous opioids by bolus, with patient- or nurse-controlled delivery systems. Although there is no doubt they have a beneficial effect on pain, opioids are associated with dose-related side effects including "over"sedation, ileus, urinary retention, nausea, vomiting, pruritus, mental confusion and respiratory depression leading to a prolonged extubation time.

In the last decades many has been written about the value of multimodal pain protocols to treat acute postoperative pain in non-cardiac surgery. This is not only to reduce the dose and side effects of opioids. By blocking both the central and peripheral pain mechanisms the aim is to find a holy grale, by which the patient suffers the least, by which central neural hyper-excitability that increases postoperative pain is minimized and by which the transformation of acute into chronic pain is reduced to a minimum.

Pregabalin has his role in treating various neuropathic pain syndromes. It inhibits central neuronal sensitization and prevents hyperalgesia by decreasing excitatory amino acid neurotransmission in the spinal cord through a direct postsynaptic or presynaptic inhibition of Ca²+ influx. It has been shown that gabapentin reduced pain scores and opioid requirements in different surgical settings. Literature is not conclusive and because of conflicting results the routine use of gabapentin and pregabalin to reduce opioid consumption in the cardiac surgical patients is not yet recommended.

Dexmedetomidine is an alpha-2 adrenergic receptor agonist that can be directly applied to the peripheral nervous system, causing a dose-dependent inhibition of C-fibers and Aα-fibers. It is widely used for sedation and anxiolysis in ICU settings. The clinical efficacy has been proven in non-cardiac surgery by augmenting anesthesia and analgesia, and allowing a reduction in opioid requirements. Additionally, there was a significantly lower incidence of postoperative delirium.

Ketamine isn't only an anesthetic agent but also has an analgesic effect. The exact mechanism is not yet known but some of the pathways are already identified. It binds to the opioid receptors κ(kappa) δ(delta) μ(mu) and it was proven that ketamine induces phosphorylation of mitogen-activated protein kinases by 2-3 times that of traditional opioid drugs. Another way of producing its analgesic effect is by the muscarinic acetylcholine receptors in the central nervous system. Ketamine also effects other ion channels including sodium channels and voltage sensitive calcium channels leading to local anesthetic and gabapentin like effects. Because of the unique effect of keeping hemodynamic stability during induction, ketamine can be useful in cardiac surgery. The analgesic effect, the absence of respiratory depression and hemodynamic stability make it an excellent drug to use in the ICU.

Intravenous lidocain during the perioperative period has many beneficial effects in open procedures, such as an earlier return of gastrointestinal tract function, less postoperative opioid consumption, improvement of postoperative cognitive dysfunction and reduced stay in the hospital. The exact working mechanism isn't 100% identified but the anti-inflammatory effects of LA mediated through interactions with polymorphonuclear cells and the inhibition of G protein-coupled receptors may play a crucial role for the observed effects in the perioperative setting.

Magnesiumsulphate's analgesic mechanisms are also not fully identified, but it is thought that the NMDA (N-methyl-d-aspartate) receptor is blocked by calcium regulation mechanisms. Because the NMDA receptor plays a role in the transmission of pain, magnesium has become a subject of interest as potential use in postoperative painschemes. It was proven that peri-operative intravenous magnesium can reduce opioid consumption especially in the first 24h.

The investigator's goal is to compare standard "Fentanyl - Tramadol - Paracetamol - Oxycodon" regimen to a multimodal painmanagement "pregabalin- magnesiumsulphate - minimal fentanyl-ketamine-lidocain-dexmedetomidine- paracetamol" to determine which therapy provides the most comfort, the fastest extubation time, the least pain and the least delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first time cardiac surgery by median sternotomy
* Elective surgery or semi-urgent: there needs to be time to provide 1 hour before surgery the intake of pregabalin
* ≥ 18 years for men
* Women who are in menopause
* Possibility to communicate with the patient to score pain and comfort
* Signed Informed Consent, signed by subject able and willing to provide written informed consent for study participation

Exclusion Criteria:

* Urgent surgery
* Women who are in premenopause
* Hypersensitivity to any of the study medication
* In case of direct postoperative revision the patient is NOT excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harlinde Peperstraete, MD, Principal Investigator — UZ Gent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start on January 21, 2019, primary completion on December 1st, 2021.
Groups:
- Classical Protocol: Fentanyl Max. 15µg/kg IV Per-operative
  Ultiva (Remifentanyl) 0.02-0.1µg/kg/h IV Post-operative
  Paracetamol 4x1g /24h IV Post-operative
  Tradonal (Tramadol) 100mg IV 4/d IV Post-operative in case of break through pain
  Oxynorm (Oxycodon) 5-10mg 4-6/d PO Post-operative in case of Break through pain
- Multimodal Protocol: Lyrica (Pregabalin) 75mg PO 2 hours before the operation
  Dexdor (Dexmedetomidine) 0.8µg/kg/h IV Per-operative / Post-operative
  Ketalar (Ketamine) Bolus (0.5mg/kg) + 0.3mg/kg/h IV Per-operative until stop propofol
  Linisol (Lidocain) Bolus (1.5mg/kg) + 1.3mg/kg/h IV Per-operatiive until 12h post-op
  Magnesium Sulphate Induction (25mg/kg) + 25mg/kg weaning ECC IV Per-operative
  Fentanyl 2.5µg/kg IV Per-operative
  Paracetamol 4x1g /24u IV Post-operative
  Tradonal (Tramadol) 100mg IV 4/d IV Post-operative in case of Break through pain
  Oxynorm (Oxycodon) 5-10mg 4-6/d PO Post-operative in case of Break through pain
  Dexmedetomidine: The use of multimodal painkillers pre, per and postoperative
Period: Overall Study
Arm/Group | Classical Protocol | Multimodal Protocol
Started | 50 | 50
Completed | 50 | 46
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Classical Protocol | Multimodal Protocol | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 9 | 27
  >=65 years | 32 | 37 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (9.4) | 71.2 (8.1) | 70.7 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 41 | 38 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Belgium | 50 | 46 | 96

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain After Cardiac Surgery
Description: By using a NRS scale postoperative pain (at rest) at 48hours after cardiac surgery In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10 . Zero usually represents 'no pain at all' whereas 10 represents 'the worst pain ever possible'.
Time Frame: At 48 hours after cardiac surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Classical Protocol | Multimodal Protocol
Number analyzed (Participants) | 50 | 46
units on a scale | 2.28 (1.906) | 2.17 (2.039)

2. Secondary Outcome: (ICDSC)Delirium After Stop Sedation by Using Intensive Care Delirium Screening Checklist
Description: delirium in the direct postoperative phase, by using the ICDSC (Intensive Care Delirium Screening Checklist) score. The ICDSC is score-based (range 0-8) where the ICDSC is positive when any four (or more) symptoms of delirium are present (i.e., altered level of consciousness, inattention, disorientation, hallucinations or delusions, psychomotor activity, inappropriate speech or mood, sleep disturbance or fluctuation of symptoms)
Time Frame: At 48 h after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Classical Protocol | Multimodal Protocol
Number analyzed (Participants) | 50 | 46
score on a scale | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

ADVERSE EVENTS:
Time Frame: 7days
Arm/Group | Classical Protocol | Multimodal Protocol
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/46
Other Adverse Events (participants affected / at risk) | 0/50 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/72/NCT04987372/Prot_SAP_001.pdf